CLINICAL TRIAL: NCT01848262
Title: ECALMIST (Early CPAP And Large Volume Minimal Invasive Surfactant Therapy) Versus InSurE (Intubate, Surfactant, Extubate) in Preterm Infants With Respiratory Distress Syndrome (RDS): Prospective Randomised Control Clinical Trial
Brief Title: ECALMIST Versus InSurE in Preterm Infant < 32 Weeks,Multicenter, Multinational RCT
Acronym: ECALMIST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Yahya Al Ethawi, Dr, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2013:054
Record Dates: First submitted 2013-05-02; First posted 2013-05-07 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-02

CONDITIONS: Respiratory Distress Syndrome
Keywords: ECALMIST; InSurE; CPAP; Ventilation; Vascular Catheter
MeSH Terms: conditions — Respiratory Distress Syndrome; Respiratory Aspiration | interventions — Insure Cement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ECALMIST (Active Comparator): ECALMIST will be used in preterm infants between 24 weeks to 31 weeks in the 1st day of life with RDS and spontaneously breathing with decision to give surfactant
  Interventions: Procedure: ECALMIST
- InSurE (Experimental): InSurE will be used in preterm infants between 24 weeks to 31 weeks in the 1st day of life with RDS and spontaneously breathing with decision to give surfactant
  Interventions: Procedure: InSure

INTERVENTIONS:
Procedure: ECALMIST — Surfactant administration via 17 (5 French) gauge, 133 mm length vascular catheter. 5 ml/kg will be drawn up in a 5 or 10 ml syringe. The vascular catheter will be inserted through the vocal cords under direct vision using a standard laryngoscope with the appropriate blade for gestational age. The procedure will be done without removing the NCPAP. A bolus of surfactant of 0.25-0.5 ml will be administered, after observing the surfactant moving up and down as indication of accurate intubation of the trachea. The surfactant will be slowly injected by small pulses of 0.25-0.5 ml over 20-30 seconds, each bolus with 10 seconds apart. At the end of the procedure, the operator will flush the catheter with 0.5 ml of air before removing the catheter.
  Other Names: CPAP and Minimal Invasive Surfactant Therapy
  Arms: ECALMIST
Procedure: InSure — Patients who will receive surfactant via this technique will have their NCPAP removed and then they will be orally intubated with a standard endotracheal tube (ETT) using standard endotracheal intubation procedures using appropriate size ETT according to the birth weight. Bovine surfactant will be administered through the ETT using the same technique described above for arm 1. Manual lung inflation using a Jackson -Rees anesthesia bag at 20/5-cm H2O pressure will be performed during the surfactant instillation after which the patient will be extubated promptly as per the discretion of the neonatal team. Immediately following extubation, nCPAP support will be recommenced. No premedication, such as sedation or atropine, will be used during either procedure.
  Other Names: Intubate surfcatant extubate
  Arms: InSurE

SUMMARY:
Minimally invasive surfactant therapy via a small vascular catheter - ECALMIST (Early CPAP And Large Volume Minimal Invasive Surfactant Therapy) versus InSurE (Intubate, Surfactant Extubate) in preterm infants with Respiratory Distress Syndrome (RDS): A prospective randomized clinical trial.

DETAILED DESCRIPTION:
After meeting all the inclusion criteria, eligible infants will be randomized to receive surfactant either through the ECALMIST or the InSurE methods. The attending neonatologist or neonatal team will have full discretion to decide when to intubate and when to extubate or wean the infant off the ventilator or NCPAP.

General guidelines for reintubation include persistent pH<7.20, PaCO2 > 65 mmHg, very frequent apnea (>2-3/hour of apneic or bradycardic spells not responsive to corrective therapy), frequent desaturations >3/hour not responding to increase in FiO2 or increase in FiO2 to 100%), or apneas requiring prolonged PPV. For the purpose of the study a successful outcome for the primary objective will have occurred if the infant has not been reintubated and ventilated during the initial 3 days of life.

ELIGIBILITY:
Inclusion Criteria:

All should apply:

* Newborn less than 32 weeks gestation at birth
* Postnatal age < 24 hrs of life
* Clinical diagnosis of RDS
* Spontaneously breathing on NCPAP
* Clinical decision to give surfactant.

Exclusion Criteria:

* Lack of parental consent.
* Need for mechanical ventilation
* Major congenital malformation

Ages: 24 Weeks to 31 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of early ventilation hours | 3 days
  The number of the newborn infants needed ventilation in the 1st 3 days of life

SECONDARY OUTCOMES:
Apnea | 15 minutes
  Pause or stop of breathing for more than 20 seconds or stop of breathing that associated with decrease oxygen saturation below 75% or decrease heart rate below 100 during ECALMIST or InSurE method of surfactant therapy
Bradycardia | 15 minutes
  Decreased heart rate below 100 beat per minutes during ECALMIST or InSurE procedure
Desaturation | 15 minutes
  Decreased level of oxygen saturation measured by pulse oximeter to below 75% for more than 20 seconds during either ECALMIST or InSurE
Total ventilation hours | hospital admition days
  Number of total hours during which the newborn are ventilated during hospital admission (form delivery till discharge home)
Incidence of Chronic lung disease | 1st 2 months of life
  The incidence of Chronic lung disease (CLD) both definitions; the need for oxygen support at 28 days of postnatal life and at the 36 weeks of corrected postnatal age
Early ventilation hours | 3 days
  The mean of ventilation hours

OTHER OUTCOMES:
Hospital stay | 1st three months of life
  The number of days that newborn spent in the hospital after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Yahya Ethawi, MD, Principal Investigator — University of Manitoba
Locations (2):
- Canada (2):
  - Health sciences Center, Winnipeg, Manitoba
  - St Boniface Hospital, Winnipeg, Manitoba